CLINICAL TRIAL: NCT06845501
Title: PURICA : Purine Supplementation in Patients With AICA-Ribosiduria
Brief Title: Purine Supplementation in Patients With AICA-Ribosiduria
Acronym: PURICA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: University Hospital of Saint-Etienne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 24CH171; 2024-A02001-46 (Other: ANSM)
Record Dates: First submitted 2025-02-20; First posted 2025-02-25 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: AICA-ribosiduria Due to ATIC Deficiency
Keywords: AICA-Ribosiduria; ATIC; purine

STUDY DESIGN:
Intervention Model Description: prospective, N-of-1 trial, comparative before/after study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Individual with AICA-ribosiduria due to ATIC deficiency (Experimental): Individual with AICA-ribosiduria due to ATIC deficiency
  Interventions: Dietary Supplement: purine-rich diet

INTERVENTIONS:
Dietary Supplement: purine-rich diet — diet to achieve a purine intake of 160mg/d

SUMMARY:
AICA-Ribosiduria due to ATIC deficiency is a rare genetic metabolic disease that affects less than 10 patients (PMID: 32557644). It results in severe polyhandicap linked to neurodevelopmental disorders, visual impairment, growth retardation, severe spinal deformities and scoliosis, and often early-onset epilepsy. The disease is caused by dysfunction of the ATIC enzyme, which is involved in de novo purine biosynthesis. A recent study (PMID: 38244287) reported a decrease in disease biomarkers in a single patient after 3 months on a purine-rich diet, which persisted for at least 1 year. The investigators propose to replicate this study on several patients to investigate the potential of this treatment for this severe orphan disease.

ELIGIBILITY:
Inclusion Criteria:

* Individual affected by AICA-ribosiduria due to ATIC deficiency

Exclusion Criteria:

- Individual already on a purine-rich diet theoretical contraindication to a purine-rich diet

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-04-24 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
Urinary concentration | 6 months
  Urinary concentration of AICA-Riboside and Succinyladenoside in mmol/mol (same unit for both).

SECONDARY OUTCOMES:
Number of hospitalizations | 12 months
  Comparison of the number of hospitalizations per time unit during the 12 months preceding the introduction of treatment, and during periods when at least one of the biomarkers has a value below 50% of the baseline (considering that these periods correspond to treatment at an effective dose and duration).
Quality of life score | 6 months
  Measurement of quality of life scores before treatment, at the end of the first phase of treatment before elimination, and at the end of the study. Tool: standardised paediatric PedsQL parent-proxy scale (a scale designed to assess the overall impact on quality of life of a paediatric patient's health status, as reported by their parents, consisting of 23 questions rated from 0 to 5 and where higher scores indicate better quality of life). In the case of adult patients, the Short Form-36 scale is used, consisting of 36 questions divided into 8 dimensions (and with a score ranging from 0 to 100). Each question is evaluated on a Likert scale, with 3, 5 or 6 possible levels of response. The 8 dimensions are also used to calculate two individual quality of life scores: the Physical Composite Score (PCS) and the Mental Composite Score (MCS). The higher the score, the greater the ability.

CONTACTS AND LOCATIONS:
Overall Officials: Francis RAMOND, doctor of medicine, Principal Investigator — Centre Hospitalier Universitaire de Saint Etienne
Locations (1):
- Chu Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No
For the moment, only one French center is conducting this study.